CLINICAL TRIAL: NCT03535779
Title: Characterisation of Human B Cell Maturation in Response to Vaccination
Acronym: BVAC
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Principal Investigator, Lucy Garvey, Consultant HIV/GU Medicine, Imperial College Healthcare NHS Trust
Other Study IDs: 16SM3542
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines; Hepatitis B Surface Antigens; Tetanus Toxoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Healthy volunteers receiving Tetanus (Td/IVP) vaccine were enrolled onto the study for 1 month with no additional follow up visits.
  Interventions: Biological: Tetanus Toxoid
- Group 2: Healthy volunteers receiving the Hepatitis B (HBsAg) vaccine were enrolled onto the study for 2 months with no additional follow up visits.
  Interventions: Biological: Hepatitis B

INTERVENTIONS:
Biological: Hepatitis B — The Hepatitis B virus, is a double stranded DNA virus that prevents Hepatitis B in the population
  Other Names: HBsAg
  Groups: Group 2
Biological: Tetanus Toxoid — The Tetanus vaccine, also known as tetanus toxoid (Td/IVP), is an inactive vaccine used to prevent tetanus in the population
  Other Names: Td/IVP
  Groups: Group 1

SUMMARY:
This study is an exploratory single site sample collection study at St Mary's hospital campus, Imperial College London. Sixteen participants scheduled to receive routine immunizations for Td/IPV (group 1) and HBsAg (group 2) will be recruited overall. Eights participants will be allocated to group 1 and eights participants to group 2 depending on their immunisation regime.

DETAILED DESCRIPTION:
The aim of the study is to characterise the maturation of human B cell response to immunization with vaccines (HBsAg and Td/IPV) known to induce long-term memory responses.

The primary objective is to characterize the number and phenotype of memory B cells induced by routine vaccination. These responses will be used as a comparison to those currently induced in HIV-1 vaccination trials.

The development of an effective HIV-1 vaccine is highly dependent on our understanding of the immune response to HIV-1 infection/vaccination. It is generally accepted that the generation of long-lived neutralising memory B cell antibody responses will be critical for an effective vaccine against HIV-1. Successful vaccines are capable of inducing long-lived B cell memory that can maintain antibodies for decades, typical examples being those induced by Hepatitis B (HBsAg) and tetanus vaccination which generates antibodies with a half-life of greater than 5 years. In contrast, current HIV-1 vaccination typically induces a short-lived B cell response with antibodies waning within a half-life of 6 months. Recent observations have shown that vaccination does not produce a homogenous population of memory B cell but rather a constellation of subsets depending on the type of vaccination.

Investigators are only beginning to understand the varying and important roles of some of these elusive subsets. Therefore understanding potential differential responses of these memory B cell subsets to successful licensed vaccines may prove critical in the creation of novel, effective vaccines to HIV-1.

The field has been energised in recent years by the identification of different memory B cell subsets. Four of these subsets can be characterised through differential expression of surface markers CD27, IgD and IgM, typically: CD27+IgD+IgM+ B cells, CD27+IgD-IgM+ B cells, CD27+IgD+IgM- B cells and CD27+IgD-IgM- IgG+/IgA+/IgE+ B cells (Mroczek ES et al, Front Immunol. 2014;5:96). Understanding how HBsAg and tetanus (as part of the Td/IPV vaccine) modulates antigen specific responses across these four memory B cell subsets will help define how Investigators understand the establishment of long-term immunological memory and may help us understand how Investigators can induce such memory responses with new HIV vaccine candidates. Data from these studies will be used to compare responses elicited by HIV vaccines in current phase I studies and determine potential defects in the maturation of vaccine induced memory.

Investigators therefore wish to obtain blood draws from individuals undergoing routine HBsAg and Td/IPV vaccination. This will allow us to isolate memory B cells circulating in the peripheral blood and characterise the different memory B cell subsets induced by effective licensed vaccines and compare responses to those induced by current HIV-1 vaccination trials, for which Investigators already have samples banked.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers aged between 18 and 55 years scheduled to receive routine vaccination for HBsAg or booster immunisation with Td/IPV
2. Previously naïve to HBsAg vaccination
3. Available for the duration of the study
4. Willing and able to give written informed consent

Exclusion Criteria:

1. Is currently participating in another clinical trial with an investigational or non-investigational drug or device
2. Unable to read and/or speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent
3. Unlikely to comply with protocol
4. Has a condition which in the opinion of the investigator is not suitable for participation in the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy and male and female volunteers aged between 18 and 55 years old.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Memory B Cells | 12 months
  The primary endpoint will measure the proportion responding B cells in one of four memory B cell subsets (defined by differential expression of CD27, IgD and IgM markers) raised in response to HBsAg and Td/IPV vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Lucy Garvey, Paddington, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: 1 year from when the study was officially closed